CLINICAL TRIAL: NCT07404865
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Telitacicept in Adult Participants With Active Primary Sjögren's Disease
Brief Title: Phase 3 Study of Telitacicept in Active Primary Sjögren's Disease
Acronym: UPSTREAM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC18G007; pSD (Registry Identifier: Active Primary Sjögren's Disease); Telitacicept (Other: Vor Biopharma Inc.); UPSTREAM (Other: Vor Biopharma Inc.)
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Primary Sjogren's Disease
Keywords: Sjögren's Disease; pSD; Primary Sjogren's Syndrome; Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental): Telitacicept
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — Subcutaneous injection
  Other Names: RC18; RC18-L
  Arms: Telitacicept
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
Phase 3 Study of Telitacicept in Active Primary Sjögren's Disease (UPSTREAM)

DETAILED DESCRIPTION:
Telitacicept (RC18) is a recombinant fusion protein designed to target B-cell-mediated immune pathways. It consists of the extracellular domain of transmembrane activator and calcium modulator and cyclophilin ligand interactor (TACI) linked to the Fc portion of human immunoglobulin G1 (IgG1).

Telitacicept binds with high affinity to the cytokines B-lymphocyte stimulator (BLyS, also known as BAFF) and A Proliferation-Inducing Ligand (APRIL). By binding these soluble factors, telitacicept prevents their interaction with cell-surface receptors on B cells, including TACI, B-cell maturation antigen (BCMA), and BAFF receptor (BAFF-R).

This inhibition reduces BLyS/APRIL signaling, leading to decreased B-cell survival, reduced differentiation of B cells into immunoglobulin-producing plasma cells, and lowering of autoantibody production, increased BLyS and APRIL levels, B-cell hyperactivity, and autoantibody production are associated with multiple autoimmune diseases.

Modulation of the BLyS/APRIL pathway is intended to reduce pathogenic B-cell activity and downstream immune effects that contribute to disease manifestations in Sjogren's disease and other B-cell-mediated autoimmune conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years of age (both inclusive) at screening
2. Participants must meet the 2016 American College of Rheumatology (ACR)/EULAR classification criteria for primary Sjogren's Syndrome at the time of screening.
3. ESSDAI ≥5 at screening (score calculated excluding renal, pulmonary and neurological domains)
4. Participants are seropositive for antibodies to Sjogren's Syndrome A (SSA)/Anti-Sjogren's Syndrome A (Ro) at the Screening Visit.

Additional inclusion criteria are defined in the protocol

Exclusion Criteria:

1. Participants who have a systemic autoimmune disease other than Primary Sjogren's Disease, such as rheumatoid arthritis, systemic lupus erythematosus, or systemic sclerosis, that can better explain the majority of the symptoms (i.e., secondary Sjogren's Disease)
2. Participants who have another autoimmune disease or inflammatory condition that could interfere with assessment of response of Primary Sjogren's Disease to therapy (e.g., systemic sclerosis, inflammatory bowel disease, gout).
3. Participants with severe fibromyalgia that could interfere with the assessment of response of Primary Sjogren's Disease to therapy
4. Active life-threatening or organ-threatening complications of Primary Sjogren's Disease at the time of screening based on investigator evaluation
5. Significant, uncontrolled medical disease in any organ system not related to Primary Sjogren's Disease (e.g., poorly controlled asthma, cardiovascular disease, accelerated hypertension, major depression, etc.) that in the opinion of the investigator would preclude participant participation.

Additional exclusion criteria are defined in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of telitacicept versus placebo at Week 48 in the change from baseline in the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score at Week 48. | Week 48
  Change from baseline in the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score at Week 48.

SECONDARY OUTCOMES:
To evaluate the efficacy of telitacicept versus placebo at Week 48 in the treatment of adult participants with pSD. | Week 48
  To evaluate the efficacy of telitacicept versus placebo at Week 48 in the treatment of adult participants with pSD.
To evaluate the efficacy of telitacicept versus placebo in improving glandular function during the trial. | Week 48
  Change from baseline in the stimulated whole salivary flow at Week 48.
To evaluate the effect of telitacicept versus placebo in improving patient-reported outcomes (i.e., how participants feel and function) during the trial. | Week 48
  Change from baseline in the EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) score at Week 48
To evaluate the efficacy of telitacicept versus placebo at Week 48 in the change from baseline in the physician's global assessment of disease activity (Physician GDA) score at Week 48 | Week 48
  Change from baseline in the physician's global assessment of disease activity (Physician GDA) score at Week 48
To evaluate the efficacy of telitacicept versus placebo at Week 48 in the change from baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) score at Week 48 | Week 48
  Change from baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) score at Week 48
To evaluate the efficacy of telitacicept versus placebo at Week 48 in the change from baseline in the participant's global assessment of disease activity (Patient GDA) at Week 48. | Week 48
  Change from baseline in the participant's global assessment of disease activity (Patient GDA) at Week 48.

IPD SHARING:
Plan to Share IPD: No